CLINICAL TRIAL: NCT01293383
Title: A Phase 1 Study Evaluating the Safety of LEO 90105 and Its Vehicle, After Multiple Administration on Intact Skin of Healthy Japanese Male Subjects. A Single Centre, Prospective, Randomised, Double-blinded, Vehicle-controlled Clinical Study
Brief Title: A Study Evaluating the Safety of LEO 90105 and Its Vehicle, After Multiple Administration on Intact Skin of Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MCB 0902
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 90105 (Other)
  Interventions: Drug: LEO 90105
- Vehicle (Other)
  Interventions: Drug: LEO 90105

INTERVENTIONS:
Drug: LEO 90105 — Ointment

SUMMARY:
The purpose of this trial is to to investigate the safety of LEO 90105 compared with its vehicle after multiple administration (twice daily, 5 days) in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects
* Aged 20 to 40 years inclusive
* Subjects without signs of skin irritation (erythema, dryness, roughness or scaling) on the test site
* Subjects willing to follow the study procedures and complete the study
* Subjects having understood and signed a written informed consent
* Subjects without abnormal in physiological test and clinical test in screening, and also judged as possible to participant the study by investigators

Exclusion Criteria:

* Subjects with Body mass Index (BMI ) (body weight(kg)/height (m)²) outside the range 18-25 kg/m2(18≤BMI<25)
* Subjects with history of alcohol, chemical or drug abuse
* Subjects with history of allergic reaction to any content of the study medication
* Subjects with systemic or cutaneous disease that could in any way confound interpretation of the study results (e.g. atopic dermatitis, eczema, psoriasis)
* Subjects with known sensitivity to any component of any of the formulations being tested
* Subjects with known hepatic, renal or cardiac disorders
* Subjects using systemic, locally injected or inhaled corticosteroids within 4 weeks of study start (Day 1)
* Subjects using systemic vitamin D analogues,vitamin D or calcium supplements within 4 weeks of study start (Day 1)
* Subjects using any drug (systemic or topical) within 2 weeks of study start (Day 1)
* Subjects using non-marketed/other investigational products one month prior to or 5 half lives (for those the half life is longer than one month) and during the trial is not permitted
* Subjects with any abnormality found at medical interview before administration of the test drug, which will affect the clinical study as judged by the investigator
* Subjects with history of or active photo-induced or photo-aggravated disease (abnormal response to the sun light)
* Subjects with exposure to excessive or chronic ultraviolet (UV) radiation i.e., sunbathing, tanning salon use, phototherapy) within four weeks prior to study start (Day 1) or planned during the study period
* Subjects with scars, moles, sunburn, or other blemishes in the test area which would interfere with grading
* Subjects whose partner wishes to become pregnant but is unwilling to use birth control during the study
* Subjects with any condition which, in the opinion of the investigator, would place the subject at an unacceptable risk if he participated in the study
* Subjects with any disease which are contradictions for treatment of the investigation products or for which treatment with the investigation products needs to be carefully considered (Subjects with any of the following conditions present on the area(s) to be treated with study medication: viral (e.g., herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers or wounds)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Skin irritation | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Masanari Shiramoto, MD., PhD, Principal Investigator — Hakata Clinic LTA Clinical Pharmacology Center
Locations (1):
- Hakata Clinic LTA Clinical Pharmacology Center, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en